CLINICAL TRIAL: NCT06204783
Title: Real-time Pressure Volume Loop Monitoring as a Guide for Enhanced Understanding of Changes in Elemental Cardiovascular Physiology During Therapeutic Strategies Aiming for Hemodynamic Optimization. Cohort II: Structural Heart Interventions (PLUTO-II)
Acronym: PLUTO-II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Nicolas van Mieghem, prof. dr. N.M. Van Mieghem, Erasmus Medical Center
Other Study IDs: PLUTO-II
Record Dates: First submitted 2023-02-13; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure; Valvular Heart Disease; Aortic Stenosis; Mitral Insufficiency; Tricuspid Insufficiency
Keywords: Pressure-volume loop; Cardiac mechanoenergetics
MeSH Terms: conditions — Heart Failure; Heart Valve Diseases; Aortic Valve Stenosis; Mitral Valve Insufficiency; Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort A: Transaortic Valve Implantation (TAVI): Elective TAVI with biventricular PV loop monitoring (throughout the procedure)
  Interventions: Other: Pressure volume (PV) loop measurement
- Cohort B: Mitral Transcatheter Edge-to-Edge Repair (mitral TEER): Elective mitral TEER with biventricular PV loop monitoring (throughout the procedure)
  Interventions: Other: Pressure volume (PV) loop measurement
- Cohort C: Tricuspid Transcatheter Edge-to-Edge Repair (tricuspid TEER): Elective tricuspid TEER with biventricular PV loop monitoring (throughout the procedure)
  Interventions: Other: Pressure volume (PV) loop measurement

INTERVENTIONS:
Other: Pressure volume (PV) loop measurement — Pressure volume (PV) loop measurement using a conductance catheter

SUMMARY:
The aim of PLUTO-II is to use biventricular pressure-volume (PV) loop measurements to improve the understanding of direct changes in cardiac and hemodynamic physiology induced by transcatheter aortic valve implantation (TAVI) or tricuspid edge-to-edge repair (TEER). These procedures evoke immediate changes in cardiac mechanoenergetics, ventricular-vascular interaction as well as ventricular (in)dependency. Within the context of PLUTO-II, patients will undergo biventricular PV-loop measurements before and after TAVI or TEER. In future, the application of perprocedural PV loop monitoring may tailor the daily individual decision making process during structural interventions in the catheterization laboratory.

DETAILED DESCRIPTION:
Pressure-Volume (PV) loop monitoring is a tool allowing direct visualization of individual cardiac and hemodynamic physiology, including parameters reflecting cardiac mechanoenergetics (a derivative of the myocardial metabolic demand) as well as the ventricular-arterial coupling. The concepts of changing biventricular cardiac and hemodynamic physiology induced by structural heart interventions, including Transcatheter Aortic Valve Implantation (TAVI), Transcatheter Edge-to-Edge Mitral Repair (mitral TEER) and Transcatheter Edge-to-Edge Tricuspid Repair (tricuspid TEER) are largely based on hypotheses, computer simulations and non-invasive (echocardiographic) estimations. PVL monitoring has the potential to identify unique characteristics of TAVI, mitral TEER and tricuspid TEER from the perspective of changing baseline cardiovascular physiology, including (a change in) interference between both ventricles (i.e. the ventricular crosstalk). Perprocedural (biventricular) PV loop monitoring can be of direct clinical relevance by appreciating the ventricular tolerance of increased cardiac afterload induced by the particular intervention in individual patients. In future, real-time PV loop analysis can be adjunctive to the individual decision-making process during routine structural interventions.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients undergoing elective Transcatheter Aortic Valve Implantation (TAVI) or Transcatheter Edge-to-Edge repair (TEER).

Exclusion Criteria:

* Confirmed or suspected (concomitant) congenital heart disease.
* Mechanical circulatory support (including Impella, PulseCath, Intra-Aortic Balloon Counterpulsation or Extracorporeal Membrane Oxygenation) was used during the procedure aiming to improve native cardiac output.
* No (written) informed consent was obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective TAVI or mitral TEER.
Sampling Method: Probability Sample
Enrollment: 157 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-05-14 (Estimated); Study Completion 2025-05-14 (Estimated)

PRIMARY OUTCOMES:
Cardiac mechanoenergetics | Periprocedural time window
  The change in cardiac mechanoenergetics (stroke work, potential energy and pressure-volume area in mmHg/mL) induced by the particular procedure

SECONDARY OUTCOMES:
Stroke volume (mL) | Periprocedural change (directly before vs. after the procedure)
  Based on perprocedural conductance catheter measurements
Preload recruitable stroke work (mmHg/mL) | Periprocedural change (directly before vs. after the procedure)
  Based on perprocedural conductance catheter measurements
Tau (ms) | Periprocedural change (directly before vs. after the procedure)
  Based on perprocedural conductance catheter measurements
Intraventricular dyssynchrony (%) | Periprocedural change (directly before vs. after the procedure)
  Based on perprocedural conductance catheter measurements
dP/dt min and dP/dt max (mmHg/sec) | Periprocedural change (directly before vs. after the procedure)
  Based on perprocedural conductance catheter measurements
End-systolic elastance (Ees) and arterial elastance (Ea) (mmHg/mL) | Periprocedural change (directly before vs. after the procedure)
  With Ees/Ea ratio reflecting ventricular-vascular coupling
End-systolic and end-diastolic volume (mL) | Periprocedural change (directly before vs. after the procedure)
  Based on perprocedural conductance catheter measurements
End-systolic and end-diastolic pressure (mmHg) | Periprocedural change (directly before vs. after the procedure)
  Based on perprocedural conductance catheter measurements
Starling Contractile Index (mmHg/mL) | Periprocedural change (directly before vs. after the procedure)
  Based on perprocedural conductance catheter measurements
V0, V15, V30 and V100 mmHg (mL) | Periprocedural change (directly before vs. after the procedure)
  Based on perprocedural conductance catheter measurements
SW/PVA ratio (based on the primary outcome) | Periprocedural change (directly before vs. after the procedure)
  Based on perprocedural conductance catheter measurements
Beta (ventricular stiffness constant, unitless) | Periprocedural change (directly before vs. after the procedure)
  Based on perprocedural conductance catheter measurements
Mortality | 30-day follow-up
  All-cause
Hospital stay | 30-day follow-up
  in days
Postprocedural morbidity (%) | 30-day follow-up
  including acute kidney failure, cardiac decompensation and unexpected need for vasopressor or inotropic support (all yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas M Van Mieghem, Prof MD PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van den Enden AJM, van den Dorpel MMP, Mondellini GM, Mattace-Raso AM, Adrichem R, Bastos MB, Schreuder JJ, Lenzen MJ, Kardys I, Geleijnse ML, Nuis RJ, Daemen J, Burkhoff D, Van Mieghem NM. Immediate changes in left ventricular cardiac mechanics following transcatheter aortic valve replacement for severe aortic stenosis - an in-vivo pressure-volume analysis study. Am Heart J. 2026 Mar;293:107302. doi: 10.1016/j.ahj.2025.107302. Epub 2025 Nov 14. PMID 41241186